CLINICAL TRIAL: NCT01018355
Title: The Effect of Device Closure of Patent Foramen Ovale in Elderly Patients With Crytogenic Stoke/TCI
Acronym: CryptoCard
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dissatisfactory enrollment rate
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Christian Stevns Hansen / Dr. of medicine, Ph.d. student, Department of cardiology and endocrinology at Hillerød Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hillerod-294
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2009-11

CONDITIONS: Patent Foramen Ovale; PFO; Stroke; TIA
Keywords: Patent foramen ovale; PFO; Stroke; TIA; Percutaneus closure; Intervention
MeSH Terms: conditions — Foramen Ovale, Patent; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device closure of PFO (Experimental): Device closure of PFO followed by 6 month treatment with clopidogrel 75 mg and 75 - 150 mg of aspirin daily followed by a life long treatment with dipyridamol 200 mg twice daily plus 75-150 mg aspirin daily
  Interventions: Device: Percutaneous device closure of patent foramen ovale
- Medical anticoagulative treatment (Active Comparator): Life long treatment with dipyridamol 200 mg twice daily plus 75-150 mg aspirin daily
  Interventions: Device: Percutaneous device closure of patent foramen ovale

INTERVENTIONS:
Device: Percutaneous device closure of patent foramen ovale — Percutaneous device closure of patent foramen ovale

SUMMARY:
The primary objective is to evaluate if patent foramen ovale (PFO) closure and antiplatelet medical management can reduce the risk of recurrent stroke or transient ischemic attack (TIA) when compared to antiplatelet medical management alone in elderly patients above 50 years of age with a PFO and a history of cryptogenic stroke or TIA.

DETAILED DESCRIPTION:
Prior to birth the fetal heart has a connection between the two atrias of the heart. After labour this connection often closes. About 10-15 % these connections remains open. This phenomenon is called patent foramen ovale or PFO, and is in most cases unsymptomatic.

The prevalence of PFO in patients with crytogenic (without known causes) stroke is much higher (about 40%)than the general population (about 10%). This has led to the theory that the presence of PFO can lead to stroke, by the passage of emboli from the peripheral venous circulation through the PFO to the brain by right-to-left shunting of the blood.

There are no existing data from prospective randomized studies focusing on the effect of device closure PFO in patients with cryptogenic stroke. Some observational retrospective studies have shown a beneficial effect in the reduction of recurrent stoke in patients younger that 50 years with cryptogenic stroke when PFO has been closed with a percutaneous device closure(PCD). Some studies have reported an 0% to 3.4% annual recurrence rate of stroke or TIA in patients treated with PDC. The recurrence rate of stroke or TIA in patients with crytogenic stroke or TIA in ordinary antithrombotic treatment is about 5-15 %.

The primary objective of this study is to assess whether percutaneous device closure of patent foramen ovale is superior to conventional antithrombotic treatment in preventing stroke recurrence in elderly patients above 50 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Stroke or TIA within 30 days
* Above 50 years of age

Exclusion Criteria:

* Deceases og the esophagus
* Dementia
* Allergy to aspirin
* Risk of non-compliance
* Lacking ability to give written or oral consent
* Atrial Fibrillation
* Neurological deficit lasting less than 6 hours

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-09 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint defined by the time from intervention to either fatal og non-fatal stroke/TIA | Endpoints assessed every half year starting 1 year after intervention

SECONDARY OUTCOMES:
ct-verified stroke 2 years after intervention | 2 years after intervention
Death by other causes than Stroke | Endpoint assessed every half year starting 1 year after intervention
Examination of residual cardiac right to left shunt after device closure of PFO | 1 month after intervention
Complications to device closure of PFO | few days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Hansen, dr., Principal Investigator — Hillerød Hospital. dept. of cardiology and endocrinology; Niels Tønder, Dr., Study Director — Hillerød Hospital. dept. of cardiology and endocrinology; Kasper K Iversen, Dr., Study Director — Hillerød Hospital. dept. of cardiology and endocrinology
Locations (1):
- Dept. of cardiology and endocrinology H, Hillerød, Region H, Denmark